CLINICAL TRIAL: NCT06769711
Title: The Comparison of Tunnel Morphology and Graft Healing in Anterior Cruciate Ligament Reconstructions Using Peroneus Longus And Hamstring Tendons
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Fevzi Gurkan Aslan, Dr, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24237859510
Record Dates: First submitted 2025-01-01; First posted 2025-01-10 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: anterior cruciate ligament; peroneus longus tendon; hamstring tendon; snq; tunnel widening
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peroneus Longus Group (Experimental): Participants who underwent ACL reconstruction using Peroneus Longus tendon graft.
  Interventions: Procedure: Surgical procedure using Peroneus Longus for ACL reconstruction.
- Hamstring Group (Active Comparator): Participants who underwent ACL reconstruction using Hamstring tendon graft.
  Interventions: Procedure: Surgical procedure using Hamstring tendons for ACL reconstruction.

INTERVENTIONS:
Procedure: Surgical procedure using Peroneus Longus for ACL reconstruction. — Surgical procedure using Peroneus Longus for ACL reconstruction.
  Arms: Peroneus Longus Group
Procedure: Surgical procedure using Hamstring tendons for ACL reconstruction. — Surgical procedure using Hamstring tendons for ACL reconstruction.
  Arms: Hamstring Group

SUMMARY:
1. Comparison of the grafts using Magnetic Resonance Imaging (MR) to determine whether their maturation and bone integration are different,
2. Comparison of the grafts using Computerized Tomography (CT) to determine whether their effects on the tunnels opened in cruciate ligament reconstruction surgeries are different,
3. In the event that graft healing and effects on the tunnels differ between grafts, determination of whether these differences are related to patient clinics,

DETAILED DESCRIPTION:
The project method; Patients who will be operated with 2 different grafts used in anterior cruciate ligament surgeries will be included in 2 different randomized groups of 29 people (hamstring and peroneus groups) determined by obtaining their informed consent before the surgery and then,

1. The maturation of the grafts will be measured and compared with the SNQ (Signal/Noise quotient) value and the graft-bone integration with the SI (Signal Intensity) value with the Magnetic Resonance (MR) to be taken at the 1st year controls after the surgery,
2. Changes in tunnel morphology; The volume of the tunnels will be measured with the Computerized Tomography (CT) imaging method to be taken prospectively within the first week after the surgery date and 1 year after the surgery date and the changes within 1 year will be calculated by comparing them.
3. In the outpatient clinic follow-ups of both groups; Knee laxity will be obtained with Lachman, Anterior drawer and Pivot shift tests and knee scores and activity levels will be obtained using IKDC, Lysholm, Marx scales and it will be examined whether these data are related to SNQ, SI and tunnel expansion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 45 years.
* BMI in the range of 18 to 28.
* Diagnosed with an anterior cruciate ligament (ACL) injury preoperatively confirmed by MRI.
* Patients for whom it is deemed appropriate to harvest ipsilateral hamstring tendons or Peroneus Longus tendon for use as a graft.

Exclusion Criteria:

* History of previous surgery on the affected knee or ankle.
* Presence of multiple ligament injuries in the affected knee.
* Diagnosis of advanced osteoporosis.
* ACL injuries that occurred more than 12 months prior to surgery.
* Evidence of unstable meniscal injury on preoperative MRI, which may alter the postoperative rehabilitation process.
* Evidence of unstable meniscal injury on preoperative MRI, which may alter the postoperative rehabilitation process.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Graft Maturation Assessed by Signal-to-Noise Quotient (SNQ) on MRI | 1 year postoperatively.
  Comparison of graft maturation between peroneus longus and hamstring tendon autografts using SNQ values obtained from 1-year postoperative MRI.
Graft-Bone Integration Assessed by Signal Intensity (SI) on MRI | 1 year postoperatively.
  Comparison of graft-bone integration between peroneus longus and hamstring tendon autografts using SI values obtained from 1-year postoperative MRI.
Change in Tunnel Volume Assessed by CT | Within 1 week post-surgery and at 1 year post-surgery.
  Comparison of tunnel volume changes between peroneus longus and hamstring tendon autografts by measuring tunnel volume via CT imaging performed within the first week and 1 year after surgery.

SECONDARY OUTCOMES:
Knee Laxity Assessed by Clinical Tests | At 1-year follow-up.
  Comparison of knee laxity (Lachman, anterior drawer, and pivot shift tests) between groups and correlation with graft healing (SNQ, SI) and tunnel expansion.Clinical grading of laxity based on standard examination protocols.
Patient-Reported Knee Function and Activity Levels | At 1-year follow-up.
  Comparison of knee function and activity levels between groups using IKDC, Lysholm, and Marx scales and evaluation of correlations with SNQ, SI, and tunnel volume changes.Standardized scoring from IKDC, Lysholm, and Marx scales.
Relationship Between Tunnel Changes and Clinical Outcomes | At 1-year follow-up.
  Assessment of whether tunnel volume changes correlate with knee function, activity levels, or laxity test results.Statistical correlation analysis between tunnel volume changes and clinical outcomes.
Comparison of Graft Healing and Tunnel Changes Between Groups | 1 year postoperatively.
  Evaluation of whether differences in SNQ, SI, or tunnel volume changes are specific to patient demographics or clinical characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Orthopedic and Traumatology Department, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol